CLINICAL TRIAL: NCT00784901
Title: Study of the Correlation Between Macular Thickness Analyzed by Optical Coherence Tomography and the Visual Functions in Retinitis Pigmemtosa
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Muh-Shy Chen, National Taiwan University Hospital
Other Study IDs: 200807069R
Record Dates: First submitted 2008-11-02; First posted 2008-11-04 (Estimated); Last update posted 2008-11-11 (Estimated); Status verified 2008-11

CONDITIONS: Retinitis Pigmentosa
Keywords: Macular Thickness Analyzed by Optical Coherence Tomography in Retinitis Pigmemtosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Purpose: To study the associations between visual functions and the retinal tomography detected by optical coherence tomography (OCT) in patients with retinitis pigmentosa (RP).

Study design: retrospective, non-randomized and non-comparable study Material: Medical recordings of the RP patients who visited the Out-Patient Department of Ophthalmology in NTUH during June, 2003 to June, 2008.

Methods: By reviewing charts of the RP patients, the investigators will categorize RP patients into different types according to the loci of the pathological change in their retina evaluated by opththaomoscopy. And the investigators will collect the data of their visual functions including visual acuity, visual field, Arden ratio of electrooculography, and color sense discrimination. Then, according to the OCT map, the investigators will analyze the retinal thickness by dividing the macular area into foveal area, inner ring and outer ring. Finally, the investigators will analyze the relationships between visual functions and retinal thickness in different macular areas in different types of RP patients.

Anticipated results: The investigators expect that retinal tomographies may different among different types of RP. And the retinal tomographic change may correspond to the change of a certain kind of visual function. Hence, according to the thickness of a specific area in macula, the investigators may anticipate that some visual dysfunction may exist.

DETAILED DESCRIPTION:
The diagnosis of RP was according to the typical clinical history of night blindness, characteristically findings of "bone-spicule" change in the fundus, and varying degrees of peripheral visual field constriction. According to the affected loci in the fundus, we defined a typical type of RP as the retinal pathological change was around the banded area outside the main vascular arcs, and a central variant of RP stood for those with bone-spicule change appeared at the macula.[17] The exclusion criteria included eyes with histories of trauma, intraocular laser treatment, intraocular surgery, presence of retinal diseases, high degree of myopia with refraction more minus than -8.0 D or hyperopia with refraction more than +5.0 D. Patients with systemic diseases that may affect retina like diabetes or hypertension were also excluded.

Visual acuity was examined with a Snellen visual chart with a calibrated luminance. Then according to the equation that Snellen VA equals to 1/MAR (MAR= minimal angle of resolution), Snellen VA was converted into logMAR for statistics. For calculation, visual acuity of hand motion was converted into 20/2000 and light perception was converted into 20/20000 of Snellen fraction. Visula field examination was evaluated using Goldmann kinetic perimetry with varying sizes and illuminations of testing light spots. Then the degree of the widest visual field isopter was recorded. EOG: is used to assess function of retinal pigment epithelium. During dark adaptation, resting potential decreases slightly and reaches a minimum ("dark trough"). When the light is on, the resting potential increases ("light peak"). The ratio of light peak voltage versus dark trough voltage is known as the Arden ratio. The EOG was performed with pupil dilated, first in the dark for 15 minutes, and then in the light for 15 minutes and the Arden ratio for analysis was recorded.

Color sense discrimination test was evaluated using Farnsworth Munsell 100-Hue test (Munsell FM 100, X-Rite, USA). Each patient arranged four trays of colored caps in hue order. There is a predetermined sequence for each tray. The closer the patient's arrangement is to the correct sequence, the better the patient's color sense discrimination. The Farnsworth-Munsell 100-Hue Test Scoring Software was used to score the results of Farnsworth-Munsell 100-Hue Test. The results are displayed in polar or linear format, and the total error score was recorded for calculation.

OCT was performed with the ultimate commercial OCT units (OCT3, Carl Zeiss Meditec, Inc, Dublin, CA) to measure the macular thickness under papillary dilatation by an experienced examiner. The retinal thickness was calculated using OCT retinal mapping software (version 6.1 a), which measured thickness of nine divided macular regions after six scans with 6 mm long centered on the patient's fixation point by means of an inner fixation target (Figure 1), and expressed as a color-coded map. Internal fixation was essentially chosen due to better reproducibility. We defined the foveal area as the area centered at fixation with a diameter of one millimeter, the inner ring as the area between circles with diameter of one and three millimeters, and outer ring as the area between circles with diameter of three and six millimeters (Figure 2).

We analyzed and compared the patients' characteristics, results of visual function tests and macular tomography in these two groups of RP. Then we tried to find out if there were correlations between macular tomography and visual function tests

ELIGIBILITY:
Inclusion Criteria:

* Medical recordings of the RP patients who visited the Out-Patient Department of Ophthalmology in NTUH during June, 2003 to June, 2008

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Medical recordings of the RP patients who visited the Out-Patient Department of Ophthalmology in NTUH during June, 2003 to June, 2008
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muh Shy Chen, Professor, Study Chair — NTUH
Locations (1):
- Naitonal Taiwan University Hospital, Taipei, Taiwan